CLINICAL TRIAL: NCT03425578
Title: Glutamate Supplementation and Its Effects on Skeletal Muscle Glucose Metabolism During an Oral Glucose Challenge in Healthy Young Men
Brief Title: Glutamate Supplementation in Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ORE#: 22581
Record Dates: First submitted 2018-01-17; First posted 2018-02-07 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Monosodium glutamate; Amino acids; Glucose tolerance
MeSH Terms: interventions — Sodium Glutamate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSG + CHO (Experimental): Participants will ingest 150 mg/kg body mass monosodium glutamate followed by 75 g dextrose.
  Interventions: Dietary Supplement: MSG; Dietary Supplement: CHO
- MSG + placebo B (Active Comparator): Participants will ingest 150 mg/kg body mass monosodium glutamate followed by a non-caloric, flavoured placebo.
  Interventions: Dietary Supplement: MSG; Dietary Supplement: Placebo B
- Placebo A + CHO (Active Comparator): Participants will ingest placebo capsules followed by 75 g dextrose.
  Interventions: Dietary Supplement: CHO; Dietary Supplement: Placebo A

INTERVENTIONS:
Dietary Supplement: MSG — 150 mg/kg body mass monosodium glutamate (MSG).
  Arms: MSG + CHO; MSG + placebo B
Dietary Supplement: CHO — 75g CHO (i.e. dextrose)
  Arms: MSG + CHO; Placebo A + CHO
Dietary Supplement: Placebo A — A non-caloric placebo composed of table salt (NaCl) and sucralose (Splenda).
  Arms: Placebo A + CHO
Dietary Supplement: Placebo B — A non-caloric placebo composed of flavoured water.
  Arms: MSG + placebo B

SUMMARY:
Amino acids play an important role in human metabolism. In aging individuals and in some diseases, certain amino acids, such as glutamate, are at lower than normal levels. Glutamate appears to be involved in providing energy and maintaining normal blood sugar (glucose) levels, processes which both depend heavily on skeletal muscle. The maintenance of healthy blood sugar levels, in particular, is tightly related to overall muscle mass and quality. To better understand the link between glutamate and glucose metabolism in skeletal muscle, the investigators will be using a nutritional approach to raise the body's glutamate levels with monosodium glutamate (MSG) supplementation, and raise blood glucose levels with a sugary drink. By altering the normal levels of glutamate and glucose in the blood and muscle tissue, the investigators can gather more information about the role of glutamate in energy metabolism. This will help the design of future studies investigating the function of glutamate in aging and disease. During this study the investigators will increase the levels of glutamate and glucose in the bloodstream by asking participants to ingest MSG along with a sugary drink. The goal is to subsequently determine: A) the amount of glutamate and glucose that ends up in the muscle; and B) whether normal skeletal muscle glucose metabolism, and the behaviour of additional amino acids (other than glutamate) is altered. The hypothesis is that when MSG and sugar drink are ingested together glucose uptake and metabolism within the skeletal muscle will be elevated.

DETAILED DESCRIPTION:
Glutamate is involved in several aspects of glucose metabolism in both muscle and liver, however its role has not been fully defined. It is the primary amino acid taken up by resting and exercising skeletal muscle, where it interacts with pyruvate (derived from glycolysis) to produce the TCA cycle intermediate 2-oxoglutarate and the gluconeogenic precursor alanine. Glutamate is also required for the production of glutamine, another gluconeogenic precursor, via intramuscular reactions with ammonia. Given that skeletal muscle is responsible for 85% of whole body glucose disposal, investigating the interplay between glutamate, its related amino acids, and glucose homeostasis is of particular relevance. However, despite its many links to energy provision, the role of glutamate in skeletal muscle glucose metabolism remains poorly understood.

Few studies have manipulated circulating concentrations of both glutamate and glucose in humans, and none have evaluated the effect of this unique manipulation in skeletal muscle tissue. In healthy young adults, a dose of roughly 10 g monosodium glutamate (MSG) transiently elevates plasma (700-800%) and intramuscular (30%) glutamate concentrations. Acute MSG supplementation also stimulates modest increases in plasma concentrations of aspartate, alanine, and glutamine (which are produced from glutamate within the muscle and subsequently released into circulation). Intriguingly, insulin is secreted in response to MSG supplementation, an effect that appears to be mediated by glutamate binding to an excitatory amino acid receptor on the pancreas. In addition to its action on the pancreas, there is some evidence to suggest that glutamate may function as a secondary messenger by enhancing glucose-stimulated insulin secretion during periods of increased carbohydrate (CHO) availability. However this secondary effect of glutamate on insulin is poorly understood.

The ability of glutamate to independently stimulate insulin secretion provides further support for an association between glutamate and glucose metabolism, yet only two studies to date have administered MSG during an oral glucose challenge to directly examine this relationship. One study observed no effect of MSG on glucose tolerance, however peak plasma glutamate was dramatically blunted in this study compared to previous reports (~ 80 vs. 400-500 µM), likely due to glutamate being retained in the gut as a result of co-ingestion with CHO. In a separate study, the authors developed a methodological approach to circumvent this issue: by staggering the administration of MSG and CHO by 30 min, plasma glutamate and glucose were both significantly and simultaneously elevated. Furthermore, MSG administration improved glucose tolerance. In support of these findings, improvements in glucose clearance following a high-fat meal combined with MSG has also been reported. Interestingly, not all studies have observed enhanced insulin secretion with higher glutamate availability. This suggests that the ability of carbohydrate to stimulate insulin secretion may overpower any effect of glutamate on this hormone, but the specific mechanisms remain to be fully elucidated.

Recently, investigators have developed a cell culture model to show that glutamate stimulates glucose uptake in rat L6 myotubes in the absence of insulin. This suggests that glutamate is capable of acting directly on skeletal muscle, and supports previous findings of improved glucose tolerance with acute MSG supplementation despite no further increase in insulin secretion. Additionally, cell data demonstrates that glutamate-stimulated glucose uptake results from increased glucose transporter 4 (GLUT4) translocation to the sarcolemma, via the activation of AMP-activated protein kinase (AMPK) and p38 mitogen-activated protein kinase (MAPK). It is possible that these mechanisms underpin glutamate-mediated improvements in glucose tolerance in humans. However, this - as well as the fate of glucose upon being taken up by the muscle cell - has yet to be investigated.

There is a high degree of interplay between glutamate and glucose metabolism, but it remains unclear whether elevated plasma concentrations of glutamate and glucose influence one another's uptake into human skeletal muscle, as well as their subsequent respective intramuscular metabolic reactions. Therefore, the overarching goal of this study is to uncover the effects of acute MSG+CHO supplementation on plasma and intramuscular amino acid concentrations, as well as aspects of skeletal muscle glucose metabolism, in healthy young men in comparison to the ingestion of MSG and CHO alone.

The investigators will stagger the administration of MSG and CHO by 30 min to achieve simultaneous peak circulating concentrations of glutamate and glucose. Under these conditions, the aim is to:

Primary:

1. Quantify and compare changes in circulating glutamate and intramuscular glutamate following MSG+CHO versus MSG alone.
2. Evaluate the acute effects of MSG+CHO on the intramuscular free amino acid pool (specifically aspartate, alanine, and glutamine) compared with MSG adminstration alone.

Secondary:

1. Confirm the findings of our previous study (7) which demonstrated that MSG+CHO attenuates the rise in plasma glucose (but does not affect insulin or C-peptide concentrations) compared with CHO alone.
2. Determine if MSG+CHO is associated with a greater or lesser degree of signaling through the AMPK/p38 MAPK and/or insulin pathway in skeletal muscle compared to MSG and CHO alone.
3. Explore whether aspects of skeletal muscle glucose uptake, storage, and/or utilization are altered during MSG+CHO, relative to CHO alone.

The investigators hypothesize that when glutamate and glucose are simultaneously available in peak concentrations in circulation they will observe:

Primary:

1. Lower circulating and intramuscular glutamate concentrations following MSG+CHO versus MSG alone.
2. Similar intramuscular concentrations of aspartate, alanine, and glutamine in response to MSG+CHO and MSG alone.

Secondary:

1. A blunted increase in plasma glucose (but no difference in insulin or C-peptide concentrations) following MSG+CHO compared with CHO alone.
2. Elevated expression and activation of proteins related to both AMPK/p38 MAPK and insulin signaling following MSG+CHO. However, AMPK/p38 MAPK signaling will be greatest following MSG alone, with negligible activation of the insulin signaling pathway. Conversely, insulin signaling will be greatest following CHO alone, with negligible signaling through AMPK/p38 MAPK.

Enhanced skeletal muscle glucose uptake (i.e. increased GLUT4 translocation to the plasma membrane) and utilization (i.e. increased rates of glycolysis and flux through the TCA cycle), compared to the administration of CHO alone.

Eligible young men who have consented to participate will visit the laboratory on 4 occasions each separated by a washout period of approximately 1 week. Following a series of baseline assessments to evaluate body composition, fitness etc.(Visit 1), participants will complete 3 trials (Visits 2, 3 and 4) in a randomized order. For each of the 3 trials, participants will arrive by car or via public transportation at the laboratory after an 8-12 hour overnight fast (no food or drink except for water after midnight the night before). A catheter will be inserted into an antecubital vein and a fasting blood sample will be drawn (~8 mL). Participants will then consume either 150 mg/kg body mass MSG or a placebo within 5 min. Blood (~8 mL) will be drawn at the following time points: 10, 20, 30, 40, 50, 60, 75, 90, 105, and 120 min. Immediately following the 30 min blood draw, participants will consume a 75 g carbohydrate (dextrose) beverage or a second placebo. After the last blood sample is obtained the catheter will be removed. The total amount of blood drawn during each trial will be ~88 mL.

ELIGIBILITY:
Inclusion Criteria:

* BMI in the normal or overweight range (18.5-30.0 kg/m2)
* Weight stable for the past 6 months
* Participate in aerobic and/or resistance-type exercise 3-5 times per week (no more then 2 hours per session and/or 5 sessions per week)
* Fasting blood glucose < 6.0 mM
* Resting blood pressure < 140/90 mmHg
* Answer "no" to all questions on the Get Active Questionnaire (GAQ)

Exclusion Criteria:

* Smoking
* Known allergy or intolerance to MSG
* Diabetes, cancer, or other metabolic disorders
* Cardiac or gastrointestinal problems
* Infectious disease
* Injuries that prevent safe participation and exercise or instructions from healthcare provider to refrain from exercise
* Barium swallow or nuclear medicine scan in the previous 3 weeks
* If receiving a DXA scan will cause the participant to exceed the maximum trivial dose of radiation per year
* Prescription anti-coagulant or anti-platelet medication (e.g. warfarin, heparin, clopiodogrel)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Glutamate | ~ 2 hours post-ingestion
  Circulating and intramuscular concentrations by HPLC

SECONDARY OUTCOMES:
Glucose | ~ 2 hours post-ingestion
  Circulating concentrations using a spectrophotometric assay
Skeletal muscle glucose uptake | ~ 2 hours post-ingestion
  As indicated by GLUT4 and laminin co-localization (immunohistochemistry)
Insulin | ~ 2 hours post-ingestion
  Circulating concentrations using radioimmunoassay
C-peptide | ~ 2 hours post-ingestion
  Circulating concentrations using radioimmunoassay
Aspartate | ~ 2 hours post-ingestion
  Circulating and intramuscular concentrations by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Marina Mourtzakis, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibala MJ, MacLean DA, Graham TE, Saltin B. Anaplerotic processes in human skeletal muscle during brief dynamic exercise. J Physiol. 1997 Aug 1;502 ( Pt 3)(Pt 3):703-13. doi: 10.1111/j.1469-7793.1997.703bj.x. PMID 9279819
- [Background] Di Sebastiano KM, Bell KE, Barnes T, Weeraratne A, Premji T, Mourtzakis M. Glutamate supplementation is associated with improved glucose metabolism following carbohydrate ingestion in healthy males. Br J Nutr. 2013 Dec;110(12):2165-72. doi: 10.1017/S0007114513001633. Epub 2013 Jun 11. PMID 23750536
- [Background] Chevassus H, Renard E, Bertrand G, Mourand I, Puech R, Molinier N, Bockaert J, Petit P, Bringer J. Effects of oral monosodium (L)-glutamate on insulin secretion and glucose tolerance in healthy volunteers. Br J Clin Pharmacol. 2002 Jun;53(6):641-3. doi: 10.1046/j.1365-2125.2002.01596.x. PMID 12047489
- [Background] Hosaka H, Kusano M, Zai H, Kawada A, Kuribayashi S, Shimoyama Y, Nagoshi A, Maeda M, Kawamura O, Mori M. Monosodium glutamate stimulates secretion of glucagon-like peptide-1 and reduces postprandial glucose after a lipid-containing meal. Aliment Pharmacol Ther. 2012 Nov;36(9):895-903. doi: 10.1111/apt.12050. PMID 22978669
- [Background] Bertrand G, Gross R, Puech R, Loubatieres-Mariani MM, Bockaert J. Evidence for a glutamate receptor of the AMPA subtype which mediates insulin release from rat perfused pancreas. Br J Pharmacol. 1992 Jun;106(2):354-9. doi: 10.1111/j.1476-5381.1992.tb14340.x. PMID 1382779
- [Background] Bertrand G, Puech R, Loubatieres-Mariani MM, Bockaert J. Glutamate stimulates insulin secretion and improves glucose tolerance in rats. Am J Physiol. 1995 Sep;269(3 Pt 1):E551-6. doi: 10.1152/ajpendo.1995.269.3.E551. PMID 7573433
- [Background] Mourtzakis M, Graham TE. Glutamate ingestion and its effects at rest and during exercise in humans. J Appl Physiol (1985). 2002 Oct;93(4):1251-9. doi: 10.1152/japplphysiol.00111.2002. PMID 12235022
- [Background] Graham TE, MacLean DA. Ammonia and amino acid metabolism in skeletal muscle: human, rodent and canine models. Med Sci Sports Exerc. 1998 Jan;30(1):34-46. doi: 10.1097/00005768-199801000-00006. PMID 9475642
- [Background] Graham TE, Turcotte LP, Kiens B, Richter EA. Effect of endurance training on ammonia and amino acid metabolism in humans. Med Sci Sports Exerc. 1997 May;29(5):646-53. doi: 10.1097/00005768-199705000-00010. PMID 9140902
- [Background] Wagenmakers AJ. Muscle amino acid metabolism at rest and during exercise: role in human physiology and metabolism. Exerc Sport Sci Rev. 1998;26:287-314. PMID 9696993
- [Background] Graham TE, Sgro V, Friars D, Gibala MJ. Glutamate ingestion: the plasma and muscle free amino acid pools of resting humans. Am J Physiol Endocrinol Metab. 2000 Jan;278(1):E83-9. doi: 10.1152/ajpendo.2000.278.1.E83. PMID 10644540
- [Background] DeFronzo RA. Glucose intolerance and aging. Diabetes Care. 1981 Jul-Aug;4(4):493-501. doi: 10.2337/diacare.4.4.493. PMID 7049632